CLINICAL TRIAL: NCT03640208
Title: Evaluating the Effectiveness of A Proposed 11-Step Community-Based Interventional Program That Educates, Assesses Risk And Overcomes Barriers to Complete Screening Colonoscopy Among Average Risk African Americans
Brief Title: Educate, Assess Risk and Overcoming Barriers to Colorectal Screening Among African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CASE10217
Record Dates: First submitted 2018-08-14; First posted 2018-08-21 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer
Keywords: health disparities; African American; risk assessment; secondary prevention
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Complete colorectal screening (Experimental): 11 step process divided into three phases: 1. Community Outreach Event; 2. Data Collection; 3. Navigation and Program Monitoring
  Interventions: Behavioral: Education presented by trained caregiver

INTERVENTIONS:
Behavioral: Education presented by trained caregiver — After participants complete the Pre-test, an educational session will be presented by a trained caregiver, delivered in a lecture-style manner with Power Point projection of educational material. The slides in this presentation will be scripted to mitigate variability among different presenters. Topics addressed in the presentation include: CRC basics (including brief anatomy), data on disparity, risk factors, screening modalities, preventative measures, population disparities of CRC, colonoscopy exam and other screening tests. The emphasis will be on CRC risks factors and prevention. All required information that is needed to correctly answer post-test questions is embedded within the presentation.

SUMMARY:
The burden of colorectal cancer (CRC) is unequal among various populations within the United States. This inequality is most notable among African Americans, who exhibit the highest CRC mortality of all US populations. This study aims to evaluate a community-based intervention to educate, assess risk, and overcome barriers to screening among African Americans who are 45 years or older with no personal history of CRC, adenomas, or inflammatory bowel disease and have no family history of CRC.

Barriers being assessed include: Need for establishing care with primary care physician, need for financial assistance, need for reminder calls, need for transportation, need for appointment coordination, and need for education about colonoscopy preparation and procedure

DETAILED DESCRIPTION:
After reviewing the existing literature this study team believes that the proposed strategy is inherently unique, thus amenable to experimental inquiry.

The study will provide much needed data to define the extent to which the proposed multi-faceted approach may be effectively deployed to the target population. This includes the acquisition of data to evaluate the educational program, for which improvement in knowledge may be tested objectively using the study design, as well as survey and feasibility data which is pivotal for improving the strategy.

The 11 steps for completing cancer screening are listed below:

1. Demographic/Socio-economic information
2. Knowledge assessment and education
3. Risk assessment questionnaire "Am I Average Risk?"
4. Do I need screening colonoscopy?
5. Barriers to colorectal cancer screening
6. Outreach program evaluation
7. Participants data entered in REDCap database
8. Communication with primary care provider and navigator
9. Participant navigation
10. Evaluation of navigation services
11. Program monitoring

ELIGIBILITY:
Inclusion Criteria:

* Education Only: African American individuals 18 years and older.
* CRC colonoscopy screening : Average Risk African American individuals ages 45 - 75 who did not have a screening colonoscopy or other screening modality within the past10 years, have no history of CRC, adenomatous polyps or Inflammatory Bowel Disease (IBD) and no family history of colorectal cancer. This will be identified during outreach events (steps 3 and 4).
* It is important to note that this program may ultimately include all races as a community outreach event, however we will not analyze the data of non-African Americans.

Exclusion Criteria:

* African American individuals under the age of 18
* Colonoscopy within 10 years
* History of CRC, Adenoma, IBD
* Family history of CRC
* Fecal immunochemical test (FIT) within the past year
* Cologuard test within the past 3 years
* Flexible Sigmoidoscopy test within the past 5 years
* Colonography within the past 5 years

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2024-11-03 (Actual); Study Completion 2024-11-03 (Actual)

PRIMARY OUTCOMES:
Difference in paired pre-/post-test score | From baseline (week 0) to follow-up end of study (week 24)
  16 item knowledge questions, where each item is assessed as true, false, or not sure. A 25% improvement of knowledge between pre- and post-test scores will indicate an effective program

SECONDARY OUTCOMES:
Acceptability of intervention | At the end of education - 24 weeks
  Metrics (convenient, appropriate, effective, satisfaction) will be measured on a 5-point scale where the two most favorable categories (i.e. strongly agree and agree) will be considered a positive response.
Feasibility of Intervention | At the end of education - 24 weeks
  Measured by evaluating practicality or logistics of the proposed interventional program with 8 item dichotomous questionnaire.
  A 100% positive response on the questionnaire (all 8 items answered 'yes') will be considered a 'positive' questionnaire for an individual participant. If 80% of participants respond with an overall 'positive' questionnaire, the study will be considered feasible.
Fidelity of intervention | At the end of education - 24 weeks
  Number of documented deviations throughout the program.
  90% of the 11-step program needs to be followed. A 'deviation' would be defined as not adhering to one of the 11 steps.
Percentage of individuals aged 45-75 who have never had colon or rectal cancer screening | At the end of education - 24 weeks
  Percentage of individuals aged 45-75 who have never had colon or rectal cancer screening
Percentage of participants who found the Risk assessment questionnaire helpful | At the end of education - 24 weeks
  Metrics will be measured on a 5-point scale where the two most favorable categories (i.e. strongly agree and agree) will be considered a positive response.
Barriers faced to scheduling colorectal cancer screening | At the end of education - 24 weeks
  Percent of participants with barriers to receiving colorectal cancer screening.

CONTACTS AND LOCATIONS:
Overall Officials: Samir Abraksia, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States